CLINICAL TRIAL: NCT05475028
Title: Network Medicine Approaches to Classify Patients Suffering Heart Failure in Relation to Left Ventricle Ejection Fraction (HFpEF, HFmrEF, HFrEF) by Circulating CD4+ T Cell-derived DNA Methylation Signatures, Clinical Data, and Point-of-care Risk Calculators
Brief Title: Network Medicine Approaches to Classify Heart Failure With PReserved Ejection Fraction by Signatures of DNA Methylation and Point-of-carE Risk calculaTors (PRESMET)
Acronym: PRESMET
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Monaldi Hospital (Other); Federico II University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator Giuditta Benincasa, Biol.D, PhD, University of Campania Luigi Vanvitelli
Other Study IDs: UniCampania
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure, Diastolic; Heart Failure, Systolic; Pulmonary Hypertension; Atrial Fibrillation
Keywords: HFpEF; Interactome; CD4+ T cells; HFrEF; Liquid biopsy; Network Medicine
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure, Systolic; Hypertension, Pulmonary; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genomic DNA will be extracted from circulating CD4+ T cells isolated from peripheral blood of HF patients and healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF: We will recruit HFpEF (LVEF > 50%)
  Interventions: Other: RRBS
- HFrEF: We will recruit HFrEF (LVEF < 40%)
  Interventions: Other: RRBS
- Healthy controls: We will recruit volunteer blood donors
  Interventions: Other: RRBS

INTERVENTIONS:
Other: RRBS — Reduced Representation Bisulfite Sequencing

SUMMARY:
Heart failure (HF) is a syndrome, resulting from structural or functional impairment of ventricular filling or ejection of blood. Effective HF management depends on accurate and rapid diagnosis requiring assessment of symptoms and physical signs in combination with advanced and expensive imaging tools. However, several challenges arise from the traditional symptom-based diagnosis because co-morbidities of HF have similar presentations. This implies the need for a deeper knowledge of mechanistic links among genetic and epigenetic events governing the pathophysiology of HF leading to a novel molecular-based system to differentiate HF phenotypes. Now, it is emerging that the pathophysiology of HFpEF and HFrEF is different, it provides an opportunity to identify biomarker candidates that could aid in HF diagnosis and stratification between these two forms of the disease. The aim of PRESMET project is to perform liquid biopsy strategies to identify novel putative non-invasive epigenetic-sensitive biomarkers that could be used either alone or in combination with established diagnostic tests, such as natriuretic peptide, to help differentiate HFpEF from HFrEF. The Investigators will perform DNA methylation analysis on CD4+ T cells isolated from patients versus controls. Remarkably, big data generated from NGS tools will be analyzed by advanced network-oriented algorithms. Our results may provide a useful clinical roadmap in order to improve precision medicine and personalized therapy of HF.

DETAILED DESCRIPTION:
The Investigators will perform the first Network Medicine approach to integrate the DNA methylome of circulating CD4+T cells and clinical parameters in patients with HFpEF and HFrEF.

Liquid biopsy strategies will be performed to isolate PBMCs and purificate CD4+ T cells. Successivelly, genomic DNA will be extracted on columns and will be send out for RRBS.

Network-oriented algorithms will be used to analyze DNA methylation signatures and to identify specific epigenetic changes in relation to left ventricle ejection fraction.

Network-oriented DNA methylation signatures will be integrated to the H2FPEF point-of-care calculator and, then, will be validated by the use of q-RT-PCR, WB, and ELISA.

ELIGIBILITY:
Inclusion Criteria:

* HFrEF (LVEF < 40%)
* HFpEF (LVEF > 50%)

Exclusion Criteria:

* Patients with HF with a history of a reduced LVEF ≤ 40% (HFrEF) who recover LV function (LVEF ≥ 50%)
* Chronic inflammatory diseases
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population will be composed by:
  * N=20 HFpEF (LVEF > 50%)
  * N=20 HFrEF (LVEF < 40%)
  * N=20 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Percentage of differentially methylated regions (DMRs) in CD4+ T cells | 3 months
  The Investigators will identify the panel of DMRs able to distinguish HFpEF vs. HFrEF, HFpEF vs. healthy controls, and HFrEF vs. healthy controls.
Levels of differentially expressed genes in CD4+ T cells | 1 month
  The Investigators will measure the levels of gene expression of selected genes (qRT-PCR) in HFpEF vs. HFrEF, HFpEF vs. healthy controls, and HFrEF vs. healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Napoli C, Benincasa G, Donatelli F, Ambrosio G. Precision medicine in distinct heart failure phenotypes: Focus on clinical epigenetics. Am Heart J. 2020 Jun;224:113-128. doi: 10.1016/j.ahj.2020.03.007. Epub 2020 Mar 12. PMID 32361531